CLINICAL TRIAL: NCT05630326
Title: Clinical, Laboratory, and Radiological Characteristics of Urinary Tract Infections in Infants With COVID-19
Brief Title: Association Between COVID-19 and UTIs Caused by ESBL Organism in Infants
Acronym: ABCUCEOI
Status: Completed | Type: Observational
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MRC-01-22-158
Record Dates: First submitted 2022-04-07; First posted 2022-11-29 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2022-04

CONDITIONS: Renal Insufficiency
Keywords: Chronic Kidney Diseases; Acute Kidney Injury; UTIs in infants; ESBL UTIs; chronic renal failure; UTIs with COVID-19; ESBL organisms with COVID-19
MeSH Terms: conditions — Renal Insufficiency; Renal Insufficiency, Chronic; Acute Kidney Injury; Kidney Failure, Chronic | interventions — Prevalence; Restraint, Physical; Association

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ESBL UTI: all infants with UTIs caused by ESBL producing organisms
  Interventions: Other: comparing, prevalence
- Non-ESBL UTI: all infants with UTIs caused by non-ESBL producing organisms
  Interventions: Other: assessment
- ESBL UTI with COVID-19: all infants with UTIs caused by ESBL producing organisms with COVID-19 infection
  Interventions: Other: association
- ESBL UTI without COVID-19: all infants with UTIs caused by ESBL producing organisms without COVID-19 infection
  Interventions: Other: evaluation

INTERVENTIONS:
Other: comparing, prevalence — Comparing infants with UTIs caused by ESBL organism, or non ESBL organism.
  Other Names: Data on clinical and laboratory findings are reviewed from medical records for details
  Groups: ESBL UTI
Other: assessment — comparing infants with UTIs caused by ESBL organism, or non ESBL organism.
  Groups: Non-ESBL UTI
Other: association — comparing ESBLUTI with COVID-19 and ESBL UTI without COVID-19
  Groups: ESBL UTI with COVID-19
Other: evaluation — comparing ESBLUTI with COVID-19 and ESBL UTI without COVID-19
  Groups: ESBL UTI without COVID-19

SUMMARY:
Urinary tract infections (UTIs) in infants and young children are one of the most common bacterial infections, usually febrile illness without source, frequently due to Enterobacteriaceae, mainly Escherichia coli.

Multidrug-resistant organisms including extended-spectrum beta-lactamase (ESBL) producing bacteria are becoming more prevalent. Due to the risk factors of ESBL-producing organisms in community-acquired (CA)-UTIs in infants in QATAR and Arab countries are still not studied because of the limited therapeutic options. hence, the importance of this study is to get knowledge about how to decrease the rapidly increasing in ESBL- producing bacteria, in infants, and to use antibiotics in a suitable guideline.so, The aim of this retrospective case-control study is to determine the clinical manifestations, and investigations of urinary tract infections among infants and the association with COVID-19 infection, in pediatric emergency centers at Hamad General Hospital - Qatar. From 1st January 2015 till 1st January 2022.

DETAILED DESCRIPTION:
In this retrospective, case-control study investigators will include all infants (0-1 year) with UTIs who were treated at Hamad General Hospital, pediatric division- PEC Doha, Qatar, using the electronic medical records from 1st January 2015 till January 1st, 2022, diagnosed by a positive urine culture. Investigators will look for the clinical manifestations, radiological and laboratory findings, renal scarring, ESBL-organisms, prevalence, median age, gender, and ethnic background. Participants are divided into two groups: early infancy and late infancy, ESBL UTIs and non-ESBL UTIs, and upper UTIs and lower UTIs. Finally, UTIs ESBL with COVID-19 and without COVID_19.

ELIGIBILITY:
Inclusion Criteria:

* All infants with UTIs who had been treated

Exclusion Criteria:

* Patient with a mixed urine culture.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This retrospective review of electronic medical records from the pediatric division, Hamad General hospital in Doha, Qatar, will include all treated infants (0-1 years) who were diagnosed with UTI (Approximately 300 patients) between January 1, 2015, to january 1, 2022. Data collection will be done by co-investigators for all participants.
Sampling Method: Non-Probability Sample
Enrollment: 5600 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Assessment risk factors , prevalence, and the relation between ESBL UTI and COVID-19 infection of all infants with ESBL- UTIs | 1year

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alhandi Omar Helal, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad Medical Corporation, Doha, Qatar